CLINICAL TRIAL: NCT06072352
Title: A Multicenter Randomized Controlled Trial Comparing Routine Intrapartum Vulval and Perineal Cleansing Using Chlorhexidine Versus Normal Saline to Decrease Maternal and Neonatal Infection
Brief Title: Intrapartum Vulval and Perineal Cleansing Using Chlorhexidine Versus Normal Saline
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW 21-636
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Maternal Infection During Pregnancy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine acetate solution (Experimental)
  Interventions: Other: Perineal cleansing using chlorhexidine acetate solution
- Normal saline (Active Comparator)
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Perineal cleansing using chlorhexidine acetate solution — Perineal cleansing using chlorhexidine acetate solution
  Arms: Chlorhexidine acetate solution
Other: Normal saline — Perineal cleansing using normal saline
  Arms: Normal saline

SUMMARY:
Maternal infection during pregnancy is one of the leading causes of maternal mortality, accounting for 10.7% of maternal deaths worldwide (~37,000 annually). Majority of maternal infection occurs during intrapartum (36%) and postpartum (47%) period, of which the genital tract is the source of infection in 89% of intrapartum and 54% of postpartum sepsis.

Introduction of skin flora into the genital tract during vaginal examination in women with rupture of membranes or active labour may cause intrapartum and puerperal sepsis. We hypothesize intrapartum vulval and perineal cleansing before vaginal examination could reduce the chance of peripartum infection caused by introducing the skin flora to intrauterine environment.

We plan to carry out a randomized controlled trial of intrapartum vulval and perineal cleansing using chlorhexidine, compared sterile water, prior to vaginal examination during labour and its effect on maternal and neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years old
* Live singleton pregnancy
* Planned vaginal delivery
* Term in labour (after 37+0 weeks of gestation)
* Availability of GBS result at 35-37 weeks

Exclusion Criteria:

* Preterm delivery (between 24+0 to 36+6 weeks of gestation)
* Multiple pregnancy
* Presence of fever before onset of labour
* History of antibiotics use 7 days before onset of labour
* History of adverse reaction to chlorhexidine
* Planned Caesarean delivery
* Planned delivery in other units
* Women with autoimmune disease, immunodeficiency, human immunodeficiency virus or on long term steroids
* Stillbirth
* Known genital herpes
* Genital wart during pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3500 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of endometritis, wound infection, or other infection | delivery to within six weeks of delivery
  endometritis, wound infection, or other infection

IPD SHARING:
Plan to Share IPD: No